CLINICAL TRIAL: NCT00923910
Title: A Pilot Trial of WT1 Peptide-Loaded Allogeneic Dendritic Cell Vaccine and Donor Lymphocyte Infusion for WT1-Expressing Hematologic Malignancies
Brief Title: Wilm's Tumor 1 Protein Vaccine to Treat Cancers of the Blood
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Terry Fry, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 080051; 08-C-0051; NCT00608166 (obsolete NCT alias)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Results first posted 2014-05-08 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-03

CONDITIONS: Leukemia, Acute Myelogenous (AML); Leukemia, Acute Lymphocytic (ALL); Leukemia, Chronic Myelogenous (CML); Myelodysplastic Syndrome (MDS); Non-Hodgkin's Lymphoma (NHL)
Keywords: WT1 Peptide Dendritic Cell Vaccine; Hematologic Malignancies; Relapse After Allogeneic Stem Cell Transplantation; Donor Lymphocyte Infusions; WT1-Positive; Dendritic Cell Vaccine; Tumor Immunotherapy; Allogeneic Adoptive Immunotherapy; Hodgkins Lymphoma; Leukemia; Acute Myelogenous Leukemia; AML; Acute Lymphocytic Leukemia; ALL; Chronic Myelogenous Leukemia; CML; Myelodysplasia Syndrome; Non-Hodgkin Lymphoma
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin; Hematologic Neoplasms; Hodgkin Disease; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Interleukin-4; keyhole-limpet hemocyanin; Endotoxins; Diphenhydramine; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Donors (Other): Related and unrelated donors undergo lymphapheresis to prepare cellular vaccines and to donate lymphocytes for infusion.
  Interventions: Drug: Donor Lymphocytes; Drug: Diphenhydramine; Drug: Acetaminophen
- Recipients (Experimental): Participants receive donor lymphocytes and vaccines prepared from donors.
  Interventions: Drug: WT1 Peptide-Pulsed Dendritic Cells; Drug: Donor Lymphocytes; Drug: IL-4; Drug: KLH; Drug: WT1 Peptides; Drug: Endotoxin; Drug: Diphenhydramine; Drug: Acetaminophen

INTERVENTIONS:
Drug: WT1 Peptide-Pulsed Dendritic Cells
  Other Names: Wilm's Tumor 1
  Arms: Recipients
Drug: Donor Lymphocytes — Lymphocytes from donors (related or unrelated) collected via lymphapheresis.
Drug: IL-4 — water-soluble protein; this study will use GMCSF (granulocyte macrophage colony stimulating factor)/IL-4 generated monocyte derived dendritic cells
  Other Names: Interleukin-4
  Arms: Recipients
Drug: KLH — Neoantigen known to induce helper responses; will be used concurrently as a vaccine adjuvant and control antigen.
  Other Names: keyhole limpet hemocyanin
  Arms: Recipients
Drug: WT1 Peptides — dendritic cell vaccine
  Arms: Recipients
Drug: Endotoxin — Purified lipopolysaccharide prepared from E.Coli 0:113
  Arms: Recipients
Drug: Diphenhydramine — Pre-medication
  Other Names: Benadryl
Drug: Acetaminophen — Pre-medication
  Other Names: Tylenol

SUMMARY:
Background:

* Most patients with acute lymphoblastic leukemia (ALL) and many patients with acute myelogenous leukemia (AML), chronic myelogenous leukemia (CML) and non-Hodgkin's lymphoma (NHL) have a protein called Wilm's Tumor 1 (WT1) in their cancer cells. This protein is thought to be able to influence the growth of these cancers.
* A vaccine made with the WT1 protein may boost the immune system to help fight these cancers in patients whose cancer cells contain the protein.

Objectives:

* To determine the safety, effectiveness and side effects of giving the WT1 vaccine and donor white blood cells to patients with AML, ALL, CML or NHL who have previously received standard treatment and undergone stem cell transplantation.
* To determine the immune response to the WT1 vaccine and donor white blood cells in these patients and to determine if the response is related to the amount of WT1 protein in the patient's cancer cells.

Eligibility:

* Patients between 1 and 75 years of age with the blood antigen human leukocyte antigen (HLA-A2) and the WT1 cancer protein who have persistent or recurrent blood cancers after stem cell transplantation.
* The prior stem cell transplant donor must be willing to provide additional cells, which will be used to prepare the cellular vaccines and for donor lymphocyte (white blood cell) infusions.

Design:

* Patients are given the WT1 vaccine every 2 weeks for 6 weeks (weeks 0, 2, 4, 6, 8, 10). Each vaccination consists of two injections in the upper arm or thigh.
* On weeks 0, 4 and 8, patients also receive white blood cells from a donor to enhance the immune response. The cells are also given as a 15- to 30-minute infusion through a vein about 1 hour after the vaccine injection. Donor infusions are given only to patients with mild or no graft-vs-host disease resulting from their prior stem cell transplantation.
* Periodic physical examinations, blood and urine tests, scans to evaluate disease and other tests as needed are done for 12 months after enrollment in the study.

DETAILED DESCRIPTION:
Background:

* Efforts to incorporate anti-tumor immunotherapy at stages of minimal residual disease (MRD) burden are limited by profound host immune depletion associated with standard anti-cancer therapies.
* Allogeneic blood and marrow stem cell transplantation (SCT) can be curative for a number of hematologic malignancies. Part of the success of this approach is an allogeneic immunologic reaction that has been demonstrated to play a role in the eradication of residual malignant disease after transplant in certain cancers (the so called graft-versus-leukemia, GVL, or graft-versus-tumor, GVT, effect). Nonetheless, relapse remains the primary cause of treatment failure after allogeneic SCT.
* The Wilm's tumor 1 (WT1) gene product is a tumor-associated antigen that represents a potential target for immunotherapy in a wide array of cancers. WT1 is expressed in most cases of acute leukemia and in many cases of chronic myelogenous leukemia and myelodysplastic syndromes. Importantly, WT1 has limited expression in normal tissues beyond embryogenesis. This trial represents an attempt to incorporate antigen-specific immunotherapy in the setting of allogeneic adoptive cell transfer.

Objectives:

* To determine the safety, toxicity, and feasibility of donor-derived dendritic cell vaccination and donor lymphocyte infusion (DLI) after allogeneic SCT.
* To determine the frequency and severity of graft-vs.-host disease (GVHD) in patients treated with peptide-loaded donor-derived dendritic cell vaccination and donor lymphocyte infusion (DLI).
* To evaluate whether immunologic responses to WT1-specific peptides can be generated by peptide-loaded donor-derived dendritic cell vaccination and DLI after allogeneic SCT.
* To evaluate whether clinical responses to WT1-specific peptides can be generated by peptide-loaded donor-derived dendritic cell vaccination and DLI after allogeneic SCT.
* To evaluate whether immunologic and/or clinical responses may be associated with the degree of WT1 expression by malignant cells or pre-existing donor anti-WT1 immunity.

Eligibility:

* HLA-A2 plus patients may be enrolled on this trial if they have relapsed or residual disease following allogeneic SCT for a WT1 expressing hematologic malignancy.
* Donors from the previous SCT, related or unrelated, must be 5- or 6- antigen genotypic HLA-matched (single HLA-A or B locus mismatch allowed) and HLAA2 plus.

Design:

* This is a pilot study, the primary aim of which is to assess safety and feasibility of this novel vaccine strategy aimed to enhance the GVL effect after allogeneic SCT.
* Donor-derived dendritic cells prepared from peripheral blood monocytes will be loaded with a combination of three WT1-derived peptides. These peptides are each comprised of one WT1-derived oligomeric epitope known to bind to HLA-A2 and an 11-mer protein transduction epitope known to enhance peptide loading and antigen presentation.
* Patients will receive donor-derived dendritic cell vaccines every 14 days for 6 doses. Donor leukocyte infusions (DLI) will also be administered with the vaccine.
* Study endpoints will include toxicity, feasibility, antigen-specific immunity, and disease response.
* This is an exploratory pilot trial. Up to 12 patients will be treated.
* Stopping rules will take effect if excessive toxicity (e.g., GVHD) or inability to generate vaccines are observed.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion Criteria: Patient (i.e., transplant recipient)

Age greater than 1 year and less than 75 years.

One of the following Wilm's Tumor 1 (WT1)-expressing hematologic malignancies:

1. Acute lymphocytic leukemia (ALL), less than or equal to 25 percent marrow blasts.
2. Acute myelogenous leukemia (AML), less than or equal to 25 percent marrow blasts.
3. Chronic myelogenous leukemia (CML).

   * Chronic phase, recurrent after or resistant to donor lymphocyte infusion (DLI) or resistant to available abl kinase inhibitors
   * Accelerated phase, less than 20 percent marrow blasts
   * Blastic phase, less than or equal to 25 percent marrow blasts
4. Myelodysplastic syndrome (MDS), less than 20 percent marrow blasts.
5. Non-Hodgkin's lymphoma (NHL), stage 4, less than or equal to 25 percent marrow blasts.
6. Hodgkin's lymphoma (HL)
7. There will be no restriction on the volume of extramedullary disease, with the exceptions of exclusions for central nervous system involvement or progression deemed unacceptably rapid.

   WT1 expression will be confirmed by at least one of the following criteria:
   * Greater than 15 percent of malignant cells react with anti-WT1 by immunohistochemistry.
   * Positive quantitative reverse transcription polymerase chain reaction (RT-PCR) of WT1 compared with a negative control.

   Human leukocyte antigen (HLA-A2) plus (heterozygous expression is acceptable).

   Prior stem cell transplantation (SCT): Prior HLA-matched (5-6/6 antigen or 8-10/10 allele) related or unrelated allogeneic SCT required. Must be at least 42 days post-transplant, have had recovery of transplant-associated toxicity to less than grade 2, and have post-transplant donor engraftment as defined by donor chimerism greater than 50 percent (peripheral blood), neutrophil recovery to an absolute neutrophil count (ANC) greater than 500/microl independent of myeloid growth factors, and platelet recovery to greater than 20,000/microL independent of transfusion.

   Disease status: Post-transplant residual or relapsed disease. Minimal residual disease (MRD) by polymerase chain reaction (PCR) or flow cytometry is acceptable in accordance with standard disease-specific diagnostic criteria.

   Availability of previous allogeneic donor to donate cells again.

   Prior therapy: Disease-specific therapy must be stopped at least 14 days prior to protocol Cycle 1 Day 1 (C1D1) and recovery of treatment-associated toxicity to greater than grade 2 is required prior to initiation of protocol therapy. Patients may have received prior DLI, but the last dose must be at least 28 days prior to C1D1 and there must be no active graft versus host disease (GVHD) greater than grade 1 acute or extensive chronic. Systemic immunosuppression must be stopped at least 28 days prior to protocol C1D1 and there must be no active GVHD greater than grade 1 acute or extensive chronic. There is no time restriction in regard to prior intrathecal chemotherapy provided there is complete recovery from any acute toxic effects of such. Patients receiving hydroxyurea are allowed.

   Performance status of 0, 1, 2, or 3.

   Renal function: Patients must have a serum creatinine less than or equal to 1.5 times the upper limit of normal based on age-specific normal range OR a creatinine clearance greater than or equal to 60 mL/min/1.73 m^2.

   Hepatic function: Patients must have a total bilirubin less than or equal to 2.0 mg/dl and alanine aminotransferase (ALT) less than or equal to 5 times the upper limit of normal based on age- specific normal ranges.

   Ability to give informed consent. For patients less than 18 years of age, their legal guardian must give informed consent. Pediatric patients will be included in age appropriate discussion in order to obtain verbal assent.

   Recipients of unrelated donor transplants must sign a release of information form to authorize National Marrow Donor Program (NMDP) transfer of information to the National Institutes of Health (NIH).

   Subjects of childbearing or child-fathering potential must be willing to use a medically acceptable form of birth control, which includes abstinence, while they are being treated on this study.

   Inclusion Criteria: Donor

   Weight greater than or equal to 18 kg, and for unrelated donors only age greater than or equal to 18 years

   Previous HLA-matched related or unrelated allogeneic donor. Donors must be 5-6/6 antigen or 8-10/10 allele matched.

   HLA-A2 plus (heterozygous expression is acceptable).

   Adequate venous access for peripheral apheresis, or consent to use a temporary central venous catheter for apheresis.

   Donor selection will be in accordance with National Institutes of Health (NIH)/Clinical Center (CC) Department of Transfusion Medicine (DTM) criteria and, in the case of an unrelated donor, the National Marrow Donor Program (NMDP) standards. When a potentially eligible recipient of an unrelated donor product is identified, the recipient will complete an NMDP search transfer request to allow NIH NMDP staff to contact the NMDP Coordinating Center, who will, in turn, contact the donor's prior Donor Center. The NMDP Policy for Subsequent Donation Requests will be followed and the appropriate forms (Subsequent Donation Request form and Therapeutic T Cell Collection Prescription) will be submitted as required.

   Ability to give informed consent. For donors less than 18 years of age, their legal guardian must give informed consent. Pediatric donors must give verbal assent and be cleared by social work and a mental health specialist to participate.

   EXCLUSION CRITERIA:

   Exclusion Criteria: Patient

   Active graft versus host disease (GVHD) greater than grade 1 acute or extensive chronic.

   Breast feeding or pregnant females (due to risk to fetus or newborn).

   Central nervous system (CNS) malignancy by any of the following criteria:
   * Demonstration of malignant cells in the cerebrospinal fluid (CSF) in patients with leukemia or MDS as manifested by CSF white blood cell (WBC) greater than 5/microL and confirmation of CSF blasts.
   * Cranial neuropathies deemed secondary to the underlying malignancy.
   * CNS mass lesions deemed secondary to the underlying malignancy.
   * Neuroblastoma (NB): History of CNS involvement without current evidence of CNS malignancy is NOT an exclusion.

   Rapidly progressive malignancy and/or clinically significant systemic illness (e.g., severe unstable infections or organ dysfunction) that in the judgment of the PI would likely compromise the patient's ability to tolerate this therapy or interfere with the study procedures, including but not limited to a life expectancy of less than 3 months.

   High risk of inability to comply with protocol requirements as determined by principal investigator, social work, and primary team.

   Human immunodeficiency virus (HIV) infection or human T-lymphotrophic virus type 1 (HTLV-1) infection (due to associated immune suppression and decreased likelihood of developing an immune response to the vaccine and increased risk of severe infection).

   Active hepatitis B or C infection as defined by seropositive for hepatitis B surface antigen (HbSAg) or hepatitis C and elevated liver transaminases.

   Corticosteroids (dexamethasone equivalent up to 0.1 mg/kg/day) will be permitted. Topical agents and/or inhaled corticosteroids are permitted.

   Exclusion Criteria: Donor

   History of medical illness that in the estimation of the principal investigator (PI) or Department of Transfusion Medicine (DTM)/NMDP physician poses prohibitive risk to donation.

   Anemia (Hb less than 10 gm/dl) or thrombocytopenia (less than 100,000/microliter).

   Breast feeding or pregnant females (due to risk to fetus or newborn).

   High risk of inability to comply with protocol requirements as determined by the principal investigator and donor center team.

   Positive screening test for transfusion-transmissible infection in accordance with DTM or NMDP donation standards.

   Kaposi's sarcoma

Ages: 1 Year to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-02-22 (Actual); Primary Completion 2013-10-18 (Actual); Study Completion 2016-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terry J Fry, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Appelbaum FR. Graft versus leukemia (GVL) in the therapy of acute lymphoblastic leukemia (ALL). Leukemia. 1997 May;11 Suppl 4:S15-7. PMID 9179275
- [Background] Sullivan KM, Weiden PL, Storb R, Witherspoon RP, Fefer A, Fisher L, Buckner CD, Anasetti C, Appelbaum FR, Badger C, et al. Influence of acute and chronic graft-versus-host disease on relapse and survival after bone marrow transplantation from HLA-identical siblings as treatment of acute and chronic leukemia. Blood. 1989 May 1;73(6):1720-8. PMID 2653460
- [Background] Witz JP, Roeslin N, Avalos S, Morand G, Wihlm JM. [Benign tracheo-bronchial tumors. Other tumors]. Ann Chir. 1979 Oct;33(8):541-4. No abstract available. French. PMID 229756
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2008-C-0051.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Donors: Period 1 -Donor lymphocyte collection via apheresis. Period 2 -Donor cell processing for vaccine and infusion.
- Recipients: Period 1 - Vaccine and donor lymphocyte prep Period 2 - Vaccine and donor lymphocyte administration.
Period: Period 1
Arm/Group | Donors | Recipients
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Donors | Recipients
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Donors: Donor lymphocyte collection via apheresis.
- Recipients: Vaccine and donor lymphocyte prep
- Total: Total of all reporting groups
Arm/Group | Donors | Recipients | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 3 | 4
  Between 18 and 65 years | 4 | 2 | 6
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Standard Deviation); unit: years] | 21 (9.17) | 17 (3.71) | 19 (8.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 4 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10
Disease [Number; unit: participants] — ALL, acute lymphocytic leukemia; AML, acute myeloid leukemia. Population: Donors were not evaluated.
  participants
    Hodgkin: number analyzed (Participants) | 0 | 5 | 5
    Hodgkin |  | 1 | 1
    ALL: number analyzed (Participants) | 0 | 5 | 5
    ALL |  | 3 | 3
    AML: number analyzed (Participants) | 0 | 5 | 5
    AML |  | 1 | 1
Transplantation Type [Number; unit: participants] — NMA, nonmyeloablative; MA, myeloablative; MAx2, myeloablative conditioning. This is standard terminology in the transplant field and refers to pre-transplant chemotherapy/radiation doses that require stem cell rescue. Population: Donors were not evaluated.
  participants
    NMA: number analyzed (Participants) | 0 | 5 | 5
    NMA |  | 2 | 2
    MA: number analyzed (Participants) | 0 | 5 | 5
    MA |  | 2 | 2
    MA x 2: number analyzed (Participants) | 0 | 5 | 5
    MA x 2 |  | 1 | 1
Donors [Number; unit: participants] — MSD, matched sibling donor; MRD*, matched related donor. MRD* was a 10/10 matched related parent for both transplantations. the first used marrow and the second used peripheral blood stem cells.; MUD, matched unrelated donor. Population: Recipients were not evaluated.
  participants
    MSD: number analyzed (Participants) | 5 | 0 | 5
    MSD | 3 |  | 3
    MRD*: number analyzed (Participants) | 5 | 0 | 5
    MRD* | 1 |  | 1
    MUD: number analyzed (Participants) | 5 | 0 | 5
    MUD | 1 |  | 1
Conditioning Regimen [Number; unit: participants] — TBI, total body irradiation; cyclo, cyclophosphamide; etop, etoposide; HSCT, hematopoietic stem cell transplant Population: Donors were not evaluated.
  participants
    Fludarabine/cyclophosphamide: number analyzed (Participants) | 0 | 5 | 5
    Fludarabine/cyclophosphamide |  | 2 | 2
    Cyclophosphamide, TBI, thiotepa: number analyzed (Participants) | 0 | 5 | 5
    Cyclophosphamide, TBI, thiotepa |  | 1 | 1
    HSCT1:cyclo,TBI;HSCT2:busulfan, melphalan, etop: number analyzed (Participants) | 0 | 5 | 5
    HSCT1:cyclo,TBI;HSCT2:busulfan, melphalan, etop |  | 1 | 1
    Cyclophosphamide, TBI: number analyzed (Participants) | 0 | 5 | 5
    Cyclophosphamide, TBI |  | 1 | 1
Immunosuppression [Number; unit: participants] — BMT, bone marrow transplant Population: Donors were not evaluated.
  participants
    Cyclosporine: number analyzed (Participants) | 0 | 5 | 5
    Cyclosporine |  | 3 | 3
    Sirolimus/tacrolimus, methotrexate: number analyzed (Participants) | 0 | 5 | 5
    Sirolimus/tacrolimus, methotrexate |  | 1 | 1
    None after second BMT: number analyzed (Participants) | 0 | 5 | 5
    None after second BMT |  | 1 | 1
Time Off Immunosuppression before Protocol Enrollment [Number; unit: Months] — Population: Donors were not evaluated.
  Months
    Patient 1: number analyzed (Participants) | 0 | 5 | 5
    Patient 1 |  | 10 | 10
    Patient 2: number analyzed (Participants) | 0 | 5 | 5
    Patient 2 |  | 28 | 28
    Patient 3: number analyzed (Participants) | 0 | 5 | 5
    Patient 3 |  | 11 | 11
    Patient 4: number analyzed (Participants) | 0 | 5 | 5
    Patient 4 |  | 23 | 23
    Patient 5: number analyzed (Participants) | 0 | 5 | 5
    Patient 5 |  | 9 | 9
Pre-Enrollment Disease Status [Number; unit: participants] — Population: Donors were not evaluated.
  participants
    6%-8% blasts: number analyzed (Participants) | 0 | 5 | 5
    6%-8% blasts |  | 1 | 1
    Multiple 1-2cm lymph nodes: number analyzed (Participants) | 0 | 5 | 5
    Multiple 1-2cm lymph nodes |  | 1 | 1
    5%-10% blasts: number analyzed (Participants) | 0 | 5 | 5
    5%-10% blasts |  | 1 | 1
    2% blasts: number analyzed (Participants) | 0 | 5 | 5
    2% blasts |  | 1 | 1
    5% blasts: number analyzed (Participants) | 0 | 5 | 5
    5% blasts |  | 1 | 1
Time to HCT to Relapse, mo [Number; unit: Months] — Population: Donors were not evaluated.
  Months
    Patient 1: number analyzed (Participants) | 0 | 5 | 5
    Patient 1 |  | 8 | 8
    Patient 2: number analyzed (Participants) | 0 | 5 | 5
    Patient 2 |  | 1 | 1
    Patient 3: number analyzed (Participants) | 0 | 5 | 5
    Patient 3 |  | 12 | 12
    Patient 4: number analyzed (Participants) | 0 | 5 | 5
    Patient 4 |  | 11 | 11
    Patient 5: number analyzed (Participants) | 0 | 5 | 5
    Patient 5 |  | 12 | 12
Time to First Vaccine (from day 0 of HCT), mo [Number; unit: Months] — Population: Donors were not evaluated.
  Months
    Patient 1: number analyzed (Participants) | 0 | 5 | 5
    Patient 1 |  | 14 | 14
    Patient 2: number analyzed (Participants) | 0 | 5 | 5
    Patient 2 |  | 32 | 32
    Patient 3: number analyzed (Participants) | 0 | 5 | 5
    Patient 3 |  | 14 | 14
    Patient 4: number analyzed (Participants) | 0 | 5 | 5
    Patient 4 |  | 29 | 29
    Patient 5: number analyzed (Participants) | 0 | 5 | 5
    Patient 5 |  | 15 | 15

OUTCOME MEASURES:

1. Primary Outcome: Toxicity
Description: Here is the number of participants with adverse events. For details of the adverse events, see the adverse event module.
Time Frame: 21 months
Population: Only recipients were monitored for adverse events.
Measure: Number; unit: participants
Arm/Group | Recipients
Number analyzed (Participants) | 5
participants | 5

2. Primary Outcome: Number of Participants With Graft Versus Host Disease (GVHD) Greater Than or Equal to Grade 3
Description: Acute Graft versus Host Disease (GVHD) was graded by the modified Glucksberg scale. 0 = no GVHD normal, 4 = severe GVHD.
Time Frame: 28 days following completion of last vaccine and/or DLI (donor lymphocyte infusion) administration
Population: Data for the frequency and severity of GVHD was captured as an endpoint for this trial. The donor arm is not included here because they were not evaluated for this outcome measure; recipients only.
Measure: Number; unit: participants
Arm/Group | Recipients
Number analyzed (Participants) | 5
participants | 0

3. Secondary Outcome: Time to Immune Response
Description: Immune response was monitored by use of interferon gamma Enzyme-Linked Immunospot (ELISpot) and by delayed-type hypersensitivity (DTH) testing.
Time Frame: 4 to 12 weeks
Population: The donor arm is not included here because they were not evaluated for this outcome measure; recipients only.
Measure: Number; unit: Weeks
Arm/Group | Recipients
Number analyzed (Participants) | 5
Weeks
  Patient 1 | 12
  Patient 2 | NA — Not collected.
  Patient 3 | 8
  Patient 4 | 4
  Patient 5 | 3

4. Secondary Outcome: Wilm's Tumor 1 (WT1) Enzyme-Linked Immunospot (ELISpot)
Description: WT1 expression of the hematologic malignancy was confirmed by either having greater than 15% of malignant cells react with anti-WT1 by immunohistochemistry or by having a positive quantitative reverse transcription polymerase chain reaction (RT-PCR) of WT1 compared with a negative control.
Time Frame: 48 to 72 hours after placement
Population: The donor arm is not included here because they were not evaluated for this outcome measure; recipients only.
Measure: Number; unit: participants
Arm/Group | Recipients
Number analyzed (Participants) | 5
participants
  Positive | 3
  Negative | 2

5. Secondary Outcome: Wilm's Tumor (WT1) Delayed-type Hypersensitivity (DTH)
Description: WT1 expression of the hematologic malignancy was confirmed by either having greater than 15% of malignant cells react with anti-WT1 by immunohistochemistry or by having a positive quantitative reverse transcription polymerase chain reaction (RT-PCR) of WT1 compared with a negative control. DTH skin testing was performed using KLH and with a cocktail of WT1 peptides as 2 separate injections. Enzyme-Linked Immunospot (ELISpot) was performed against each peptide and was considered positive if results were at least 10 spots above background on at least 2 measurements. DTH was considered positive if there was at least .5cm induration 48 to 72 hours after placement.
Time Frame: 48 to 72 hours after placement
Population: The donor arm is not included here because they were not evaluated for this outcome measure; recipients only.
Measure: Number; unit: participants
Arm/Group | Recipients
Number analyzed (Participants) | 5
participants
  Positive | 2
  Negative | 2
  NA (Not available) | 1

6. Secondary Outcome: Keyhole Limpet Hemocyanin (KLH) Delayed-type Hypersensitivity (DTH)
Description: KLH is a neoantigen known to induce helper response was used concurrently as a vaccine adjuvant and control antigen. DTH skin testing was performed using KLH and with a cocktail of WT1 peptides as 2 separate injections. Enzyme-Linked Immunospot (ELISpot) was performed against each peptide and was considered positive if results were at least 10 spots above background on at least 2 measurements. DTH was considered positive if there was at least .5cm induration 48 to 72 hours after placement.
Time Frame: 48 to 72 hours after placement
Population: The donor arm is not included here because they were not evaluated for this outcome measure; recipients only.
Measure: Number; unit: participants
Arm/Group | Recipients
Number analyzed (Participants) | 5
participants
  Positive | 3
  Negative | 1
  NA (Not available) | 1

7. Secondary Outcome: Number of Participants With Progressive Disease
Description: Progressive disease is at least a 20% increase in the sum of the longest diameter of all target lesions (i.e. tumor response). Response criteria for acute leukemia's is worse marrow classification (i.e., M status) with at least a 50% increase in the percentage of marrow blasts, or no change in marrow classification (i.e., M status), but a 50% or greater increase in absolute peripheral blast count or extent of medullary disease
Time Frame: 4 to12 weeks
Population: The donor arm is not included here because they were not evaluated for this outcome measure; recipients only.
Measure: Number; unit: participants
Arm/Group | Recipients
Number analyzed (Participants) | 5
participants | 5

ADVERSE EVENTS:
Time Frame: 21 months
Description: Only recipients were monitored for adverse events.
Arm/Group | Recipients
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recipients (N=5)
AST, SGOT (serum glutamic oxaloacetic transaminase) - high (Metabolism and nutrition disorders) | 3 (6)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (2)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (1)
Allergy/Immunology - Other, Specify - allergy to Sorbaview (Immune system disorders) | 1 (1)
Coagulation - Other, Specify - PT, prolonged (Blood and lymphatic system disorders) | 1 (2)
Glucose (serum -high (hyperglycemia) (Metabolism and nutrition disorders) | 2 (25)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 4 (7)
Hemorrhage, pulmonary/upper respiratory: Nose (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hepatobiliary/pancreas- Other, Specify - non-alcoholic Steatoheptits (Hepatobiliary disorders) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutriphils:lung (pneumonia) (Infections and infestations) | 1 (1)
GGT (gamma-Glutamyl transpeptidase) (Metabolism and nutrition disorders) | 1 (1)
Bicarbonate, serum low (Metabolism and nutrition disorders) | 2 (2)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 1 (1)
Albumin, serum low (hypoalbuminemia) (Metabolism and nutrition disorders) | 2 (19)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Dry eye syndrome (Eye disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0x10e9/L) (General disorders) | 3 (5)
Febrile neutropenia (Infections and infestations) | 1 (1) — Fever of unknown origin without clinically or microbiologically documented infection) (ANC <1.0x10e9/L, fever >=38.5 degrees C)
Insomnia (General disorders) | 1 (1)
Iron overload (Blood and lymphatic system disorders) | 1 (1)
Magnesium, serum high (hypermagnesemia) (Metabolism and nutrition disorders) | 2 (3)
Magnesium, serum low (hypomagnesemia) (Metabolism and nutrition disorders) | 2 (7)
Nausea (Gastrointestinal disorders) | 2 (2)
Ocular/Visual - Other, Specify - Eye drainage (Eye disorders) | 1 (1)
Pain: Abdomen NOS (Gastrointestinal disorders) | 3 (3)
Pain: Eye (Eye disorders) | 1 (1)
Pain: Head/Headache (Nervous system disorders) | 2 (3)
Pain:Joint (Musculoskeletal and connective tissue disorders) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4 (11)
Rigors/chills (General disorders) | 1 (2)
Striae (Skin and subcutaneous tissue disorders) | 1 (1)
Supraventricular and nodal arrhythmia: sinus bradycardia (Cardiac disorders) | 1 (1)
Supraventricular and nodal arrhythmia: sinus tachycardia (Cardiac disorders) | 2 (2)
Sweating (diaphoresis) (General disorders) | 1 (1)
Triglyceride, serum high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 1 (3)
Uric acid, serum high (hyperuricemia) (Metabolism and nutrition disorders) | 1 (4)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1)
Vision-blurred vision (Eye disorders) | 1 (1)
Platelets-low (Blood and lymphatic system disorders) | 5 (30)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1 (3)
Phosphate, serum low (hypophosphatemia) (Metabolism and nutrition disorders) | 1 (3)
Pain: chest wall (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain: neck (Musculoskeletal and connective tissue disorders) | 1 (1)
Mood alteration:anxiety (Nervous system disorders) | 2 (2)
Pain: throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Leukocytes (total WBC) - low (Blood and lymphatic system disorders) | 4 (26)
Infection with unknown ANC:sinus (Infections and infestations) | 1 (2)
PTT (partial thromboplastin time) (Blood and lymphatic system disorders) | 2 (2)
Pruritis/itching (Skin and subcutaneous tissue disorders) | 4 (7)
ALT, SGPT (serum glutamic pyruvic transaminase) - high (Metabolism and nutrition disorders) | 3 (12)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 1 (3)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 2 (18)
Cholesterol, serum-high (hypercholesteremia) (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Hemoglobin-low (Blood and lymphatic system disorders) | 4 (14)
Infection with normal ANC or Grade 1 or 2 neutrophils:lung (pneumonia) (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils: upper airway NOS (Infections and infestations) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) - low (Blood and lymphatic system disorders) | 4 (21)
Pain:muscle (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain:pain NOS (General disorders) | 1 (3)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2 (9)
Proteinuria (Metabolism and nutrition disorders) | 1 (1)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 3 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No